CLINICAL TRIAL: NCT06311448
Title: Personalized Targeted Immunomodulation in Patients With ARDS Related to COVID19 and Future Pandemic Pathogens
Brief Title: Personalized Targeted Immunomodulation in COVID-19 ARDS
Acronym: COMODULATE
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Amsterdam UMC (Other); Leiden University Medical Center (Other); St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Henrik Endeman, Henrik Endeman, MD, PhD, Erasmus Medical Center
Other Study IDs: 10094
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome
Keywords: Immunomodulation; Tociluzimab; Biomarker; Complement inhibitors; IL-6 inhibitors; IL-1 inhibitors; JAK inhibitors
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated with immunomodulation: Adult patients with COVID-19 ARDS admitted to ICU and requiring mechanical ventilation and receiving standard of care treatment (including steroids) and single-target immunomodulation, for example Toculizimab, Anakinra, etc.
  Interventions: Drug: Single target immunomodulation
- Not treated with immunomodulation: Adult patients with COVID-19 ARDS admitted to ICU and requiring mechanical ventilation and receiving standard of care treatment (including steroids).
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Single target immunomodulation — Single target immunomodulation compromise of drugs which very specifically target cytokines, chemokines or specific receptors, which are involved in the pathofysiology of COVID-19. For instance, tociluzimab (IL-6 receptor blocker), Anakinra (IL-1 receptor blocker), Eculizimab (Complement inhibitor C5), etc.
  Groups: Treated with immunomodulation
Drug: Standard of care — Standard of care during COVID-19 pandemic including steroids.
  Groups: Not treated with immunomodulation

SUMMARY:
Rationale: In COVID19 single-targeted immunomodulation, mostly via an IL-6 receptor blocker, was used by a one-size fits all non-targeted approach. In future pandemics the same might occur. However, for individual patients, this might not yield optimal treatment.

Objectives: This project aims to identify a way to individualize and target immunomodulation, using COVID19 as a testcase for the future.

* Identify immunological pathways which are associated with outcome in C-ARDS.
* Test whether an individualized biomarker-based approach has an effect on outcome and costs when using single-target immunomodulation in C-ARDS(Tocilizumab, Anakinra, etc.).
* Explore whether other immunological pathways were present in patients with C-ARDS which could have been intervened with medication which is already available and has been described in ARDS or similar diseases.

Study type: Retrospective observational multicenter study in the Netherlands.

Study population: Adult patients (≥ 18 years) hospitalized and admitted to the ICU with COVID-19 and acute respiratory distress syndrome (ARDS) (i.e., receiving invasive mechanical ventilation) will be included.

Intervention (if applicable): Not applicable (retrospective study design).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Given the retrospective nature of the study, no burden, risks or benefits for the patient are associated with participation. The target population of this study is specific to hospitalized patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Admitted to ICU due to COVID induced moderate or severe ARDS
* Requiring mechanical ventilation

Exclusion Criteria:

- Refusing participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years or older, admitted to the ICU due to COVID-induced moderate or severe ARDS as defined by the Berlin criteria, and requiring mechanical ventilation, were eligible for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Mortality up to day 90 | From date of ICU admission up to date of hospital discharge, assessed up to 90 days.
Change in SOFA score | During the full course of ICU-admission. The length of ICU-stays varies per patient.
  Repeated measurements of SOFA scores during ICU admission will be performed on days 0, 1, 2, 7, 14, 21 and 28. SOFA scores will be compared between days and from the start to the end of ICU admission.
Ventilator free days | During the full course of ICU admission. The length of ICU-stays varies per patient.
  Number of ventilator free days
Change in biomarker values | During the full course of ICU admission. The length of ICU-stays varies per patient.
  Repeated measurements of biomarkers during ICU admission will be performed on days 0, 1, 2, 7, 14, 21 and 28. Biomarker values will be compared between days and from the start to the end of ICU-admission.
Costs of immmunomodulation | During the full course of ICU admission. The length of ICU-stays varies per patient.
  Costs of immunomodulation will be compared to the costs of dexamethason. Furthermore, we will explore whether patients who were treated with single target immunomodulation have shorter ICU length of stay and more ventilator free days, which also reduce the total costs.

CONTACTS AND LOCATIONS:
Overall Officials: H. Endeman, Dr., Principal Investigator — Erasmus Medical Centre
Locations (1):
- Erasmus Medical Centre, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available through a secure data transfer system and appropriate data transfer agreement. (The data set contains personal data.
Supporting Information: Study Protocol